CLINICAL TRIAL: NCT05258955
Title: Comparison of Anti-plaque Efficacy of Natural Honey With Chlorhexidine Mouthwash: A Randomized Controlled Trial
Brief Title: Title: Comparison of Anti-plaque Efficacy of Natural Honey With Chlorhexidine Mouthwash: A Randomized Controlled Trial
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Liaquat National Hospital & Medical College (Other)
Collaborators: Liaquat College of Medicine and Dentistry (Other)
Responsible Party: Principal Investigator, Muhammd Abid, Registrar at LCMD, Liaquat National Hospital & Medical College
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1030419MAOM
Record Dates: First submitted 2022-02-17; First posted 2022-02-28 (Actual); Last update posted 2022-02-28 (Actual); Status verified 2022-02

CONDITIONS: Dental Plaque
Keywords: Dental plaque, Honey, Chlorhexidine
MeSH Terms: conditions — Dental Plaque | interventions — chlorhexidine gluconate

STUDY DESIGN:
Intervention Model Description: The participants divided into two groups. one group will received honey based oral rinses and other group received chlorhexidine mouthwash and will evaluate the reduction of dental plaque
Who Masked: Participant
Masking Description: The mouthwash were distributed in dark color coded bottle and marked with label A and B, as to maintain masking among the the participants of the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Chlorhexidine (Active Comparator): these are the group which received chlorhexidine based preparation for plaque reduction
  Interventions: Drug: Chlorhexidine mouthwash
- Natural honey (Experimental): these group will received the honey base mouthwash and the its effect on plaque reduction will be observed in follow up visits
  Interventions: Other: Natural honey

INTERVENTIONS:
Other: Natural honey — Natural Sidr honey based mouthwash used as intervention group B (Arm Group B) for the reduction of plaque index
  Other Names: Sidr Honey
  Arms: Natural honey
Drug: Chlorhexidine mouthwash — Chlorhexidine gluconate 0.12% mouthwash is used as intervention in Group A (Arm Group A) for the comparison of plaque reduction among group A and B
  Other Names: Chlorhexidine Gluconate
  Arms: Chlorhexidine

SUMMARY:
The rationale of our study is to compare the efficacy of natural honey base preparation with other commercially available mouthwashes i.e chlorhexidine base in prevention of dental plaque formation as honey is readily available and cost effective and organic in nature. This study will help to provide the data of our community and positive result may provide a new method of oral hygiene maintenance with fewer side effects. We will be able to deliver the best anti-plaque agent.

DETAILED DESCRIPTION:
In this study, participants will assigned into 2 group those who will fulfilled the inclusion and exclusion criteria. After the informed consent, they were divided into 2 group. Group A will received Chlorhexidine mouthwash and Group B will provided with honey based mouthwash. The participant will blinded as solution will be provided in dark color bottle to mask the study. After which the baseline plaque index will be taken followed by recording plaque index on 7th, 14th, and 21st day. The statistical analysis will be done to compare the mean difference between these 2 groups

ELIGIBILITY:
Inclusion Criteria:

1. Individual aged between 18-25
2. Retained 28 number of teeth excluding wisdom teeth

Exclusion Criteria:

1. Individual with medical illness affecting oral cavity like diabetes, sjögren syndrome, crohn disease etc
2. Multiple extraction , overhang restoration, wearing any appliance
3. Periodontal problem with pocket depth more than 3mm
4. Current or recent history of antibiotic consumption
5. Noncompliance that is unable to maintain their hygiene.
6. Pan, Betel quid and any other oral habit will not be included in study

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2020-06-03 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2021-01-21 (Actual)

PRIMARY OUTCOMES:
Dental Plaque | reduction of plaque index will be assessed on 7th day, 14th day and on 21st day
  primary outcome is to assessed the reduction on plaque level among Group A and Group B

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Abid, BDS, Principal Investigator — Registrar, Periodontology Liaquat College of Medicine and Dentistry
Locations (1):
- Liaquat College of Medicine and Dentistry, Karachi, Sindh, Pakistan